CLINICAL TRIAL: NCT03159143
Title: A Phase II, Single-arm Study of Docetaxel and Oxaliplatin in Metastatic Cisplatin-resistant Transitional Cell Carcinoma of the Urinary Bladder
Brief Title: Study of Docetaxel and Oxaliplatin in Metastatic Transitional Cell Cancer (TCC) of the Urothelial Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leonard Appleman (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor-Investigator, Leonard Appleman, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 04-055
Record Dates: First submitted 2017-05-08; First posted 2017-05-18 (Actual); Results first posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Metastatic Transitional Cell Cancer of the Urothelial Tract
MeSH Terms: interventions — Docetaxel; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: This is a non-randomized Phase II trial in metastatic transitional cell cancer (TCC) of the urothelial tract.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Docetaxel and Oxaliplatin (Experimental): Docetaxel administered at a dose of 60mg/m^2 IV infusion, followed by oxaliplatin at a dose of 110mg/m^2 as a 2 hour IV infusion.
  Interventions: Drug: Docetaxel; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Docetaxel — Docetaxel (28) is a semi-synthetic taxane which blocks mitosis by preventing microtubule depolymerization. It mediates its actions by binding to a different set of microtubule-associated proteins than paclitaxel. It is administered every 3 weeks as a 30 minute infusion at doses between 60 to 75 mg/m^2.
  Other Names: Taxotere
Drug: Oxaliplatin — Alkylating antineoplastic agent. It is administered on day 1 of each cycle at a dose of 110 mg/m^2

SUMMARY:
The purpose of this non-randomized Phase II trial was to evaluate the efficacy of a combination of docetaxel and oxaliplatin in patients with metastatic transitional cell cancer (TCC) of the urothelial tract. The primary endpoint was to assess response, as defined as a 25% reduction in measurable disease per the RECIST criteria. Measurable or evaluable objective response rate, time to disease progression and survival were also assessed.

DETAILED DESCRIPTION:
This non-randomized Phase II trial was to evaluate the efficacy of a combination of docetaxel and oxaliplatin in patients with metastatic transitional cell cancer (TCC) of the urothelial tract. The primary endpoint was to assess response, as defined as a 25% reduction in measurable disease per the RECIST criteria. Measurable or evaluable objective response rate, time to disease progression and survival were also assessed.

Treatment was administered on an outpatient basis. No other concurrent therapy for malignant disease was administered. Patients received both docetaxel and oxaliplatin, IV on day 1 of each cycle. Treatment will be repeated every 21 days for up to 6 courses in the absence of disease progression, unacceptable toxicity, or treatment delay > 3 weeks.

All patients should receive antiemetics prior to treatment. An oral or IV 5-HT3 receptor antagonist in combination with a benzodiazepene and Decadron was recommended. To mitigate docetaxel associated hypersensitivity reactions, Decadron was administered at a dose of 8mg bid, 1 day prior to, the day of, and the day after administration of docetaxel (total of 3 days)

Day 1 of each cycle:

Docetaxel was administered at a dose of 60mg/m2 IV infusion, followed by oxaliplatin at a dose of 110mg/m2 as a 2 hour IV infusion. Oxaliplatin solution was further diluted in an infusion solution of 250 mL to 500 mL Dextrose 5% in Water (D5W). Oxaliplatin was be capped at a maximum BSA of 2.0

Day 2 of each cycle:

Patients received growth factor support as needed. At the discretion of the investigator, patients were treated with both white and red cell growth factors. Generally, white cell support is recommended if patients experience a febrile neutropenia with the preceeding cycle, or are over the age of 70 yrs, and thought to be at a high risk of febrile neutropenia (74-76)

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed transitional cell carcinoma of the Urothelial tract.
* Confirmed metastatic disease.
* Measurable progressive disease is required.
* 18 years of age. Because no dosing or adverse event data are currently available on the use of oxaliplatin in patients < 18 years of age, they are excluded from this study.
* Life expectancy of greater than 6 months.
* ECOG Performance status of 0-1.
* Must have received prior treatment with standard of care chemotherapy No more than 2 prior regimens of cytotoxic chemotherapy.
* No other experimental treatment, cytotoxics or radiation 4 weeks prior to enrollment.
* Patients must have acceptable organ function as defined below:

Hematopoietic: WBC > 2500/mm3 or ANC > 1500/mm3, hemoglobin > 9.0 g/dL, platelet count > 100,000/mm3 Hepatic: Bilirubin < 1.5 mg/dL, SGOT/SGPT < 2 x ULN (< 4 x ULN if liver metastases present) Renal: Creatinine < 1.8 mg/dL

* Adequate neurologic function defined as no clinically significant peripheral neuropathy, defined as any neuropathy ≤ grade 1.
* Adequate cardiovascular function defined as no active congestive heart failure, no uncontrolled angina, no myocardial infarction within the past 6 months.

Exclusion Criteria:

* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* No prior therapy with oxaliplatin is allowed.
* No history of allergic reactions attributed to the drugs used in this study or compounds of similar chemical or biologic composition.
* No history of intolerance or allergy to the antiemetics to be administered in conjunction with the study drugs (i.e., 5 HT3 antagonists).
* No concurrent other active cancer from another primary site, except squamous cell and basal cell carcinoma of the skin.
* No other serious concomitant illness will be allowed, including interstitial pneumonia, extensive and symptomatic fibrosis of the lung, uncontrolled hypertension, unstable angina, symptomatic congestive heart failure, NYHA Class III or IV, serious cardiac arrhythmia, uncontrolled diabetes mellitus or active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-12-17 (Actual); Primary Completion 2009-06-02 (Actual); Study Completion 2009-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Appleman, MD, Principal Investigator — Univesity of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel and Oxaliplatin: Docetaxel administered at a dose of 60mg/m^2 IV infusion, followed by oxaliplatin at a dose of 110mg/m^2 as a 2 hour IV infusion.
  Docetaxel: Docetaxel (28) is a semi-synthetic taxane which blocks mitosis by preventing microtubule depolymerization. It mediates its actions by binding to a different set of microtubule-associated proteins than paclitaxel. It is administered every 3 weeks as a 30 minute infusion at doses between 60 to 75 mg/m^2.
  Oxaliplatin: Alkylating antineoplastic agent. It is administered on day 1 of each cycle at a dose of 110 mg/m2
Period: Overall Study
Arm/Group | Docetaxel and Oxaliplatin
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel and Oxaliplatin
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 66.4 [39.9 to 83.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Percentage of patients who experienced a greater than or equal to a 30% reduction in measurable disease, as per the RECIST criteria.
Time Frame: Up to 4 years
Population: Patients who received between 1 and 6 cycles of oxaliplatin with docetaxel.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel and Oxaliplatin
Number analyzed (Participants) | 19
percentage of participants | 11 [3 to 31]

2. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) will be calculated as number of months from the date of first treatment to the date of disease progression or the date of death (disease-related causes) or the cut-off date.
Time Frame: Up to 4 years
Population: Patients received at least one cycle of docetaxel and oxaliplatin and were assessed for toxic effects.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel and Oxaliplatin
Number analyzed (Participants) | 22
months | 3 [0.2 to 5.8]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of patients who achieved complete response, partial response and stable disease. DCR will be calculated from the first day of the first cycle to the date of metastatic or primary tumor relapse, or last contact date, or date of death (if death comes before disease progression), or data cut-off.
Time Frame: Up to 4 years
Population: Patients who received at least one cycle of docetaxel and oxaliplatin and were assessed for toxic effects
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Docetaxel and Oxaliplatin
Number analyzed (Participants) | 22
percentage of participants | 26.3 [12 to 49]

4. Secondary Outcome: Overall Survival
Description: The overall survival will be calculated as the number of months from the date of first treatment until death or the cut-off date.
Time Frame: Up to 4 years
Population: Patients received at least one cycle of docetaxel and oxaliplatin and were assessed for toxic effects.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel and Oxaliplatin
Number analyzed (Participants) | 22
months | 7 [4.6 to 9.4]

ADVERSE EVENTS:
Arm/Group | Docetaxel and Oxaliplatin
Serious Adverse Events (participants affected / at risk) | 16/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and Oxaliplatin (N=22)
Cardiovascular/Arrhythmia - Other (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Cardiac-ischemia/infarction (Cardiac disorders) | 1
Gastric ulcer (requires radiographic or endoscopic documentation) (Gastrointestinal disorders) | 1
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Diarrhea patients with a colostomy (Gastrointestinal disorders) | 1
Dehydration (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection with ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 1
Neurology-Other (Nervous system disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Potassium, serum-low (hypokalemia) (Blood and lymphatic system disorders) | 1
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 1
Sodium, serum-low (hyponatremia) (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and Oxaliplatin (N=22)
Platelets (Blood and lymphatic system disorders) | 3
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 7
Hemoglobin (Blood and lymphatic system disorders) | 12
Hypotension (Cardiac disorders) | 2
Insomnia (General disorders) | 2
Weight loss (General disorders) | 2
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 3
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 3
Dehydration (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 5
Anorexia (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 11
Edema: limb (Blood and lymphatic system disorders) | 5
Alkaline phosphatase (Metabolism and nutrition disorders) | 2
Neurology - Other (Specify, __) (Nervous system disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 12
Pain, Bone (General disorders) | 2
Pain, Extremity-limb (General disorders) | 2
Pain, Joint (General disorders) | 2
Pain, Vagina (General disorders) | 2
Pain, Back (General disorders) | 3
Pain, Muscle (General disorders) | 3
Pain, Abdomen NOS (General disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 2
Phlebitis (including superficial thrombosis) (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No